CLINICAL TRIAL: NCT00474591
Title: Fondaparinux Compared With Heparin to Prevent Thrombotic Complications and Graft Failure in Patients Undergoing Coronary Artery Bypass Graft Surgery
Brief Title: Fondaparinux to Prevent Thrombotic Complications and Graft Failure in Patients Undergoing Coronary Artery Bypass Graft Surgery: The Fonda CABG Study
Acronym: Fonda CABG
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: GlaxoSmithKline (Industry)
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 06-361
Record Dates: First submitted 2007-05-16; First posted 2007-05-17 (Estimated); Last update posted 2007-05-28 (Estimated); Status verified 2007-05

CONDITIONS: Coronary Bypass Graft Failure/Occlusion
Keywords: Coronary artery bypass surgery, fondaparinux, graft patency, graft occlusion, graft failure, anticoagulation
MeSH Terms: conditions — Bites and Stings | interventions — Fondaparinux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Fondaparinux

SUMMARY:
(i) Main Research Question(s): What is the effect of fondaparinux on coronary graft patency, heart attack, stroke, and death in patients who have undergone coronary artery bypass grafting (CABG)? To reliably answer this question requires a large randomised trial. We propose a pilot study to demonstrate the feasibility of recruiting patients into this study and of performing CT angiograms to measure graft patency at 30 days.

(ii) Why is this research important? Coronary artery bypass surgery has made a very important contribution to improving the health and survival of patients with advanced coronary artery disease but still has many problems. One in 10 patients experiences a heart attack at the time of surgery, 1 in 20 experiences a heart attack, stroke, or death during hospitalization, and 1 in 4 patients has at least 1 blocked graft within 1 year of surgery. Fondaparinux, a relatively new anticoagulant drug, has been shown to significantly reduce cardiovascular events and death in patients who have suffered a recent heart attack. Compared to established anticoagulant therapies for acute myocardial infarction, fondaparinux has been shown to be more effective with similar or lower risks of bleeding.

Fondaparinux, unlike the most commonly used anticoagulants, does not cause Heparin Induced Thrombocytopenia (HIT), a rare condition with extremely high morbidity and mortality.

This drug has never been studied in CABG patients. Our pilot study will provide key information about feasibility that will help us to design and perform a large definitive study in the future.

(iii) What is being studied? We will be looking at blood flow in bypass grafts, heart attack, stroke, venous thromboembolism and death. For safety we will be looking at bleeding, transfusion, and need for further surgery because of bleeding. We will also perform laboratory tests for HIT antibodies as their levels are prognostic for the development of HIT and are also related to morbidity and mortality. The incidence of actual HIT cases will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* age at least 18 years
* undergoing first ever multivessel CABG-only surgery with at least 2 free grafts (e.g. Radial artery, saphenous vein, free internal mammary artery)
* undergoing CABG with cardiopulmonary bypass

Exclusion Criteria:

* clear indication for anticoagulation (e.g. prosthetic heart valve replacement, recurrent DVT)
* allergy or intolerance of fondaparinux or unfractionated heparin
* renal failure or other contraindication for coronary artery graft CT angiogram
* inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)

PRIMARY OUTCOMES:
Graft patency | 28 days

SECONDARY OUTCOMES:
Myocardial infarction | In-hospital
Stroke | In-hospital
Death | In-hospital
Bleeding events | In-hospital, 28 days
Transfusion requirements | In-hospital
Re-operation | In-hospital

CONTACTS AND LOCATIONS:
Overall Officials: Jack CJ Sun, MD, Principal Investigator — McMaster University; John W Eikelboom, MD,MSc, Study Director — McMaster University; Kevin HT Teoh, MD,MSc, Study Chair — McMaster University; Salim Yusuf, MD,DPhil, Study Chair — McMaster University
Locations (1):
- Hamilton General Hospital, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Warkentin TE, Sheppard JI, Sun JC, Jung H, Eikelboom JW. Anti-PF4/heparin antibodies and venous graft occlusion in postcoronary artery bypass surgery patients randomized to postoperative unfractionated heparin or fondaparinux thromboprophylaxis. J Thromb Haemost. 2013 Feb;11(2):253-60. doi: 10.1111/jth.12098. PMID 23216710